CLINICAL TRIAL: NCT00709761
Title: LPT 111111- A Single-arm, Multicenter Phase II Study to Evaluate The Combination of Weekly Nanoparticle Albumin Bound Paclitaxel (Nab-Paclitaxel or ABRAXANE®) and Lapatinib (TYKERB®) in Women With No More Than One Prior Treatment for ErbB2 Overexpressing Metastatic Breast Cancer
Brief Title: Phase II Lapatinib Plus Nab-Paclitaxel As First And Second Line Therapy In her2+ MBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: LPT111111
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms, Breast
Keywords: Erbb2; ABRAXANE; MBC; first or second line therapy; Metastatic Breast Cancer; TYKERB
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Single arm combination therapy of Lap and NabPaclitaxel combination
  Interventions: Drug: Lapatinib/nab-Paclitaxel

INTERVENTIONS:
Drug: Lapatinib/nab-Paclitaxel — This was an open-label, single-arm, multi-center, Phase II study to determine the activity of nab-paclitaxel plus lapatinib (TYKERB) in the first and second-line setting in women with ErbB2 overexpressing metastatic breast cancer (MBC). Subjects were to receive nab-paclitaxel (100 mg/m2 intravenously on Day 1, 8, 15, every 28 days (q28) days plus lapatinib (1000 mg once daily on a continuous basis).

SUMMARY:
This was an open-label, single-arm, multi-center, Phase II study to determine the activity of nab-paclitaxel plus lapatinib in the first and second-line setting in women with ErbB2 overexpressing metastatic breast cancer (MBC). Sixty subjects were to be enrolled in the study. Subjects were to receive nab-paclitaxel (100 mg/m2 intravenously once weekly for 3 weeks, followed by a rest week in a 4-week cycle) plus lapatinib (1000 mg once daily). Subjects were to receive treatment until disease progression or withdrawal from the study. The primary objective of this study was to evaluate overall tumor response rate of lapatinib in combination with nab-paclitaxel administered in women with ErbB2 overexpressing MBC who received no chemotherapeutic regimen in the metastatic setting. Secondary objectives included progression-free survival, overall survival, duration of response, time to response and time to progression and safety. Safety and efficacy assessments were to be performed at 8 and 12 week intervals, and at the end of treatment.

Subject: Metastatic Breast Cancer, ErbB2, First-line therapy, Lapatinib, Nab-paclitaxel

ELIGIBILITY:
Inclusion Criteria:

A subject was eligible for inclusion in this study only if all of the following criteria apply:

* Subjects must have histologically confirmed invasive breast cancer with Stage IV disease at primary diagnosis or at relapse after curative-intent surgery. Where the disease was restricted to a solitary lesion, the neoplastic nature of the lesion should have been confirmed by cytology or histology.
* Documented amplification of ErbB2 3+ by immunohistochemistry or a positive score (>2.2) by FISH using a local laboratory result (which was considered sufficient in this study with no further verification by a central laboratory).
* Subjects must have received no more than one prior chemotherapeutic regimen in the metastatic setting.
* If a taxane had been administered in the neoadjuvant, adjuvant or metastatic setting, progression must have occurred ≥12 months after completion of this treatment.
* Prior therapy with radiation for this breast cancer population was permitted if it was administered in the neoadjuvant or adjuvant non metastatic setting. Radiotherapy given in the metastatic setting, prior to initiation of study medication, was allowed to a limited area (e.g., palliative therapy and involving less than 25% of bone marrow), if it was not the sole site of disease. Subjects must have completed radiation treatment and recovered from all acute radiation treatment related toxicities (e.g., bone marrow suppression) prior to commencement of combination treatment.
* The subject must have received all prior chemotherapy treatment at least 4 weeks prior to enrollment in this study and must have recovered from all related toxicities. Subjects who have received weekly dose of prior chemotherapy e.g. gemcitabine or capecitabine may enroll 2 to 3 weeks after cessation of treatment provided that they have recovered from all related toxicities.
* Prior therapy with trastuzumab in the neoadjuvant, adjuvant or metastatic setting was permitted. The subject must have received all prior trastuzumab treatment at least 4 weeks prior to enrollment in this study and must have recovered from all related toxicities.
* Prior endocrine therapy was permitted in the neoadjuvant or adjuvant or metastatic setting. The subject must have received all prior endocrine treatment at least 1 week prior to enrollment in this study and must have recovered from all related toxicities.
* Prior diagnosis of cancer was allowed as long as the subject was free of disease for 5 years. Subjects with completely resected basal or squamous cell skin cancer, thyroid cancer or successfully treated cervical carcinoma in-situ were allowed if it had been 1 year or greater since definitive surgery.
* Subjects must have had measurable disease, according to Response Evaluation Criteria in Solid Tumors (RECIST) guidelines; defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter [LD] to be recorded) by mammogram, ultrasound or physical exam [Therasse, 2000].
* Subjects with liver metastases or stable chronic liver disease were permitted into the study.
* Women ≥18 years of age:
* Non-child-bearing potential (i.e., women with functioning ovaries who had a current documented tubal ligation or hysterectomy, or women who were postmenopausal); or
* Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category included women with oligomenorrhoea (severe), women who were perimenopausal and young women who had begun to menstruate. These subjects must provided a negative serum pregnancy test at Screening and agree to 1 of the following:
* Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 5 days after the final dose of study medication; or
* Consistent and correct use of one of the following acceptable methods of birth control:
* Male partner who was sterile prior to the female subject's entry into the study and was the sole sexual partner for that female subject.
* Implants of levonorgestrel.
* Injectable progestogen.
* Any intrauterine device with a documented failure rate of less than 1% per year.
* Oral contraceptives (either combined or progestogen only).
* Barrier methods, including diaphragm or condom with a spermicide.
* Considered by the Investigator to have a life expectancy of ≥6 months.
* ECOG Performance Status (PS) of 0 or 1 (Karnofsky ≥80%) [Oken, 1982].
* Subjects must have had normal organ and marrow function as below:
* Hematologic
* Absolute neutrophil count ≥1.5 × 10^9/L
* Hemoglobin ≥9 g/dL
* Platelets ≥100 × 10^9/L
* Hepatic
* Serum bilirubin ≤ upper limit of normal (ULN)
* Aspartate aminotransferase ≤3 × ULN without liver metastases and alanine aminotransferase ≤5 × ULN if documented liver metastases
* Renal
* Serum creatinine ≤1.5 mg/dL
* OR -
* Calculated creatinine clearance ≥40 mL/min
* Subjects must have had a cardiac ejection fraction of >50% as measured by echocardiogram (ECHO) or multigated acquisition scan (MUGA) and within the institutional range of normal.
* Subjects with stable central nervous system metastases (stable for at least 3 months) as confirmed by computerized tomography (CT)/magnetic resonance imaging (MRI) or evidence of leptomeningeal involvement were eligible only if they were not taking steroids or enzyme-inducing anticonvulsants.
* Subject must have been free of gastrointestinal diseases that impede swallowing and retaining of oral medications.
* Signed, informed consent prior to registration.
* Bisphosphonate therapy for bone metastases was allowed; however, treatment must be initiated prior to the first dose of study medication. Prophylactic use of bisphosphonates in subjects without bone disease, except for the treatment of osteoporosis, was not permitted.
* Subjects whose disease was estrogen receptor + and/or progesterone receptor + or unknown status were included in the study if they met the following criteria:
* They had symptomatic visceral disease that required chemotherapy.
* Significant visceral organ tumor burden
* The disease was considered by the Investigator to be progressing rapidly or life threatening.
* Subjects who have received prior endocrine therapy and who were no longer benefiting from this therapy.

Exclusion Criteria:

A subject was not be eligible for inclusion in this study if any of the following criteria apply:

* Subjects who received more than one prior chemotherapeutic regimen in the metastatic setting
* Subjects taking treatment with medications provided in the list of restricted medications and substances in the drug information section for lapatinib were not eligible for the study. This included human immunodeficiency virus-positive subjects receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with lapatinib.
* Prior treatment with lapatinib.
* Concurrent anticancer or concomitant radiotherapy treatment;
* Concurrent treatment with prohibited medications;
* Use of an investigational drug within 30 days or 5 half-lives, whichever was longer, preceding the first dose of investigational treatment, or, concurrent treatment with an investigational agent or participation in another clinical trial involving investigational agents.
* Known history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or nab-paclitaxel or excipients;
* Known history of uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would have limited compliance with study requirements.
* Had active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Concurrent disease or condition that would make the subject inappropriate for study participation or any serious medical disorder that would interfere with the subject's safety.
* Pregnant or lactating females at any time during the study (due to the potential teratogenic or abortifacient effects of lapatinib and breastfeeding).
* Subjects with diseases affecting gastrointestinal function resulting in an inability to take oral medication, including; malabsorption syndrome, a requirement for iv alimentation, prior surgical procedures affecting absorption e.g. gastric resection and uncontrolled inflammatory bowel disease (e.g., Crohn's, ulcerative colitis).
* Peripheral neuropathy of Grade 2 or greater.
* Unresolved or unstable, serious toxicity from prior administration of another investigational drug and/or of prior cancer treatment.
* History of prior malignancy. However, subjects who had been disease-free for 5 years, or subjects with completely resected basal or squamous cell skin cancer, thyroid cancer or successfully treated cervical carcinoma in situ were eligible if it had been at least 1 year since definitive surgery.
* or rendering of informed consent.

Other Eligibility Criteria Considerations:

* To assess any potential impact on subject eligibility with regard to safety, the Investigator must refer to the following document(s) for detailed information regarding warnings, precautions, contraindications, AEs, and other significant data pertaining to the investigational product(s) being used in this study: Clinical Investigator's Brochure (IB), SPM, and the nab-paclitaxel Product Label.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07-02 (Actual); Primary Completion 2011-01-05 (Actual); Study Completion 2018-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (13):
  - Novartis Investigative Site, La Verne, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Salem, Virginia
  - Novartis Investigative Site, Everett, Washington
  - Novartis Investigative Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Background] Yardley DA, Hart L, Bosserman L, Salleh MN, Waterhouse DM, Hagan MK, Richards P, DeSilvio ML, Mahoney JM, Nagarwala Y. Phase II study evaluating lapatinib in combination with nab-paclitaxel in HER2-overexpressing metastatic breast cancer patients who have received no more than one prior chemotherapeutic regimen. Breast Cancer Res Treat. 2013 Jan;137(2):457-64. doi: 10.1007/s10549-012-2341-9. Epub 2012 Dec 8. PMID 23224144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Summary of subject disposition table is on the intent-to-treat (ITT) population. The ITT population comprised of all subjects who received at least 1 dose of investigational product. The ITT population, which is the same as the actually treated population, is used for all the analyses of EOS reporting.
Pre-assignment Details: A safety cohort was designed into the study to include the first 10 participants enrolled. Enrollment was halted after the enrollment of the fifth participant to allow for the safety review. Enrollment was resumed after the review and protocol amended.
Groups:
- Lapatinib 1000 mg + Nab-Paclitaxel: Participants received Lapatinib 1000 milligram (mg) tablets orally daily 1 hour before or after a meal along with a Nab-paclitaxel infusion at a dose of 100 mg/ m^2 intravenously over 30 minutes on Day 1, 8, and 15, in a 4-week cycle, for at least 6 cycles.
Period: Overall Study
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Started | 60
Completed | 33
Not Completed | 27
Not completed — Withdrawal by Subject | 8
Not completed — study closed/terminated | 17
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population comprised of all subjects who received at least 1 dose of investigational product.
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (12.78)
Age, Customized [Count of Participants; unit: Participants] — Age Group Breakdown (ITT)
  Participants
    <18 | 0
    18-64 years | 44
    65-84 years | 16
    85+ | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 50
  African American/African Heritage (Her.) | 6
  Asian | 1
  Japanese/East Asian Her./South East Asian Her. | 1
  Native Hawaiian of other Pacific Islander | 1
  American Indian of Alaska Native and White | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Tumor Response (OR)
Description: OR was defined as the percentage of participants experiencing either a confirmed complete response (CR) or a confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.0. CR is defined as the disappearance of all lesions (target and/or non-target). PR is defined as at least a 30% decrease in the sum of the longest dimensions (LD) of target lesions taking as a reference the baseline sum LD, with non-target lesions not increased or absent.
Time Frame: Start of treatment to disease progression or death or discontinuation from study or at least 28 days after last dose (up to Week 131)
Population: Intent-to-Treat (ITT) Population: all participants who received at least one dose of investigational product
Measure: Number; unit: percentage of participants
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 60
percentage of participants | 53
Statistical Analysis 1: Comparison: Lapatinib 1000 mg + Nab-Paclitaxel; Test type: Superiority or Other; percentage of participants = 53.0, 95% CI [40.7 to 66.0] — The estimation parameter represents the percentage of participants experiencing either a CR or a PR

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of treatment until death due to any cause. For participants who did not die, time to death was censored at the time of last contact. OS could not be analyzed because only 13 participants had died as of data cut off, and data were not mature (greater than 75% of the participants were censored for the endpoint).
Time Frame: Start of treatment to death (up to Week 131)
Population: ITT Population
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined for the subset of participants who showed a confirmed CR or PR, as the time from first documented evidence of CR or PR until the first documented sign of disease progression or death.
Time Frame: First documented response (CR or PR) to disease progression or death (up to Week 131)
Population: ITT Population. Only those participants experiencing a CR or a PR were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 32
weeks | 48.7 [31.7 to 57.1]

4. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined for the subset of participants who showed a confirmed CR or PR, as the time from the start of treatment until the first documented evidence of CR or PR (whichever status was recorded first).
Time Frame: Start of treatment to first documented response (CR or PR) (up to Week 131)
Population: ITT Population. Only those participants experiencing a CR or a PR were analyzed.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 32
weeks | 7.8 [7.4 to 8.1]

5. Secondary Outcome: Time to Progression (TTP)
Description: TTP was defined as the interval between the start of treatment until the earliest date of disease progression or death due to breast cancer.
Time Frame: Start of treatment to disease progression or death (up to Week 131)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 60
weeks | 41.0 [39.1 to 64.6]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the start of treatment until the earliest date of disease progression or death due to any cause, if sooner.
Time Frame: Start of treatment to disease progression or death (up to Week 131)
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Lapatinib 1000 mg + Nab-Paclitaxel
Number analyzed (Participants) | 60
weeks | 39.7 [34.1 to 63.9]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious AEs were collected from the first study drug dose administration until 30 days after the last dose and recorded on the eCRF, a total period of approximately 9.5 years.
Groups:
- Lapatinib (1000mg) + + Nab-Pacl: Participants received Lapatinib 1000 milligram (mg) tablets orally daily hour before or after a meal along with a Nabpaclitaxel infusion at a dose of 100 milligrams/meters squared (mg/ m^2) on Days 1, 8, and 15, and then every 28 days (q28), intravenously (IV) over 30 minutes weekly, in a 4 week cycle.
Arm/Group | Lapatinib (1000mg) + + Nab-Pacl
All-Cause Mortality (participants affected / at risk) | 3/60
Serious Adverse Events (participants affected / at risk) | 21/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (1000mg) + + Nab-Pacl (N=60)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Left ventricular dysfunction (Cardiac disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 1
Disease progression (General disorders) | 1
Sudden death (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Nail bed infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Ejection fraction decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lapatinib (1000mg) + + Nab-Pacl (N=60)
Anaemia (Blood and lymphatic system disorders) | 21
Leukopenia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 22
Lacrimation increased (Eye disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 53
Dyspepsia (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 39
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 23
Asthenia (General disorders) | 8
Fatigue (General disorders) | 41
Mucosal inflammation (General disorders) | 8
Oedema peripheral (General disorders) | 16
Pain (General disorders) | 5
Pyrexia (General disorders) | 11
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Haemoglobin decreased (Investigations) | 5
Weight decreased (Investigations) | 11
Decreased appetite (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11
Cognitive disorder (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 10
Headache (Nervous system disorders) | 5
Hypoaesthesia (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 23
Paraesthesia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 11
Dysuria (Renal and urinary disorders) | 4
Vulvovaginal dryness (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Acne (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 24
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 8
Nail disorder (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 29
Skin fissures (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 5
Hypotension (Vascular disorders) | 7
Lymphoedema (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.